CLINICAL TRIAL: NCT00506142
Title: A Phase 2 Study of Marqibo in Patients With Metastatic Uveal Melanoma
Brief Title: Safety and Efficacy of Marqibo in Metastatic Malignant Uveal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HBS408 (formerly IST401)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Malignant Uveal Melanoma
MeSH Terms: interventions — Vincristine

STUDY DESIGN:
Intervention Model Description: Patients were enrolled into the study in two cohorts. After completion of enrollment in Cohort 1, enrollment in Cohort 2 has commenced.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Cohort 1 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every 2 weeks.
  Interventions: Drug: Marqibo® (vincristine sulfate liposomes injection)
- Cohort 2 (Experimental): Cohort 2 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every week.
  Interventions: Drug: Marqibo® (vincristine sulfate liposomes injection)

INTERVENTIONS:
Drug: Marqibo® (vincristine sulfate liposomes injection) — Cohort 1 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every 2 weeks.
  Cohort 2 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every week.

SUMMARY:
Marqibo (liposomal vincristine) is a form of vincristine preparation. Vincristine is designed to interfere with the multiplication of cancer cells, which may slow or stop their growing and spreading throughout the body. This may cause the cancer cells to die. Liposomal vincristine is formed when vincristine is placed inside of oil droplets called liposomes, which may help to improve the delivery of drug to the tumor site. The liposomal formulation results in a slow, steady release of vincristine in the tumor metastasis, exposing the cancer cells to vincristine continuously.

The goal of this clinical research study is to learn if Marqibo (liposomal vincristine) can help to control metastatic uveal melanoma. The safety of liposomal vincristine will also be studied.

Approximately 50 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

* Uveal melanoma with histologic or cytologic confirmation of metastatic disease.
* One unidimensionally measurable lesion. If this is a cutaneous lesion it must be at least 10 mm by caliper measure. If it is a visceral or nodal or soft tissue lesion, it must be >20 mm with conventional techniques or >10 mm with spiral CT scan. Bone lesions are not considered measurable.
* Must not have received any prior systemic chemotherapy, immunotherapy, vaccine or hepatic arterial chemotherapy for metastatic disease.
* Adequate liver, renal, and bone marrow function.
* Zubrod performance status of 0-2.
* Sign an informed consent form.

Exclusion Criteria:

* Major surgery within 4 weeks of enrollment.
* Advanced symptomatic central nervous system (CNS) involvement by melanoma and those on phenytoin or requiring steroids for brain metastases, spinal cord compression, or meningeal "carcinomatosis".
* History of neurological disorders unrelated to chemotherapy (including familial neurological diseases and acquired demyelinating disorders).
* Grade 2 or greater sensory, motor and/or autonomic neuropathy at screening from any cause.
* Receiving treatment with drugs known to inhibit or induce hepatic drug metabolism by cytochrome P450-3A4 isoenzymes and/or P-glycoprotein within 1 week of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Sanders, MD, Principal Investigator — MD Anderson
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado, Denver, Denver, Colorado
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Bedikian AY, Silverman JA, Papadopoulos NE, Kim KB, Hagey AE, Vardeleon A, Hwu WJ, Homsi J, Davies M, Hwu P. Pharmacokinetics and safety of Marqibo (vincristine sulfate liposomes injection) in cancer patients with impaired liver function. J Clin Pharmacol. 2011 Aug;51(8):1205-12. doi: 10.1177/0091270010381499. Epub 2010 Oct 26. PMID 20978276

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 35 | 19
Completed | 0 | 0
Not Completed | 35 | 19
Not completed — Adverse Event | 8 | 7
Not completed — Lack of Efficacy | 21 | 7
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Physician Decision | 1 | 0
Not completed — New health condition | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Cohort 1 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every 2 weeks.
  Marqibo® (vincristine sulfate liposomes injection): Cohort 1 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every 2 weeks.
  Cohort 2 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every week.
- Cohort 2: Cohort 2 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every week
  Marqibo® (vincristine sulfate liposomes injection): Cohort 1 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every 2 weeks.
  Cohort 2 subjects will receive MARQIBO at a dose of 2.25 mg/m2 IV over 1 hour every week.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 35 | 19 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (11.43) | 66.6 (7.97) | 63.4 (10.53)
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 0 | 0 | 0
  30-59 years | 13 | 3 | 16
  >=60 years | 22 | 16 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 9 | 36
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 19 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 18 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Proportion of patients whose best overall response is complete response (CR), partial response (PR), or stable disease (SD)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 35 | 19
Participants | 18 | 8

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 15/35 | 9/19
Other Adverse Events (participants affected / at risk) | 35/35 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=35) | Cohort 2 (N=19)
ILEUS (Gastrointestinal disorders) | 2 (2) | 1 (1)
DISEASE PROGRESSION (General disorders) | 1 (1) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 2 (2)
DEATH (General disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 0 (0)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CENTRAL LINE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
KLEBSIELLA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=35) | Cohort 2 (N=19)
ANAEMIA (Blood and lymphatic system disorders) | 9 (15) | 4 (9)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (4) | 2 (3)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 2 (2)
EAR PAIN (Ear and labyrinth disorders) | 3 (3) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 2 (2) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 2 (2)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 (4) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 (15) | 7 (7)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 5 (5)
CONSTIPATION (Gastrointestinal disorders) | 25 (36) | 13 (17)
DIARRHOEA (Gastrointestinal disorders) | 16 (22) | 5 (6)
DRY MOUTH (Gastrointestinal disorders) | 1 (1) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 5 (7) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 2 (3) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 21 (39) | 10 (12)
REGURGITATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 17 (29) | 9 (13)
ASTHENIA (General disorders) | 2 (4) | 4 (5)
CHEST DISCOMFORT (General disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 6 (11) | 3 (3)
FATIGUE (General disorders) | 26 (38) | 14 (23)
FEELING OF BODY TEMPERATURE CHANGE (General disorders) | 1 (1) | 1 (1)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 4 (4) | 1 (2)
OEDEMA (General disorders) | 2 (2) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 3 (4)
PAIN (General disorders) | 12 (13) | 4 (5)
PYREXIA (General disorders) | 16 (30) | 5 (7)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 4 (8) | 2 (4)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 3 (3) | 0 (0)
FUNGAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SKIN CANDIDA (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 4 (15)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 6 (16)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (8) | 3 (6)
BLOOD CHLORIDE DECREASED (Investigations) | 0 (0) | 1 (1)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 4 (4) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 2 (4)
WEIGHT DECREASED (Investigations) | 7 (8) | 2 (2)
ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 22 (29) | 10 (10)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 7 (12) | 6 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (14) | 5 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (9) | 5 (12)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 (14) | 2 (2)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
DIZZINESS (Nervous system disorders) | 2 (2) | 3 (3)
DYSARTHRIA (Nervous system disorders) | 4 (4) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 4 (4) | 0 (0)
HEADACHE (Nervous system disorders) | 13 (14) | 6 (9)
HYPERAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 3 (4)
HYPOREFLEXIA (Nervous system disorders) | 0 (0) | 5 (10)
NEURALGIA (Nervous system disorders) | 1 (1) | 1 (3)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 15 (28) | 1 (3)
PARAESTHESIA (Nervous system disorders) | 8 (13) | 9 (19)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 8 (17) | 5 (8)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 11 (19) | 9 (23)
ANXIETY (Psychiatric disorders) | 3 (4) | 2 (4)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (3) | 0 (0)
INSOMNIA (Psychiatric disorders) | 9 (10) | 6 (6)
MOOD ALTERED (Psychiatric disorders) | 1 (1) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 13 (18) | 4 (6)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VOCAL CORD ATROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 (15) | 1 (2)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 10 (12) | 1 (2)
RASH (Skin and subcutaneous tissue disorders) | 9 (15) | 2 (4)
HOT FLUSH (Vascular disorders) | 3 (3) | 1 (1)
HYPERTENSION (Vascular disorders) | 2 (2) | 2 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 2 (2)
VASOCONSTRICTION (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No